CLINICAL TRIAL: NCT06667856
Title: Investigation of the Effectiveness of Foot Core Exercise Training with Telerehabilitation in Individuals with Rheumatoid Arthritis: a Randomized Controlled Single-Blind Study
Brief Title: Foot Core Exercise Training with Telerehabilitation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Zülal TATAR, Researcher, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Foot Core Exercise Training
Record Dates: First submitted 2024-10-24; First posted 2024-10-31 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-10

CONDITIONS: Rheumatoid Arthritis; Foot Core; Exercise
MeSH Terms: conditions — Arthritis, Rheumatoid; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Asynchronous telerehabilitation group (Active Comparator)
  Interventions: Other: Asynchronous exercise group
- Synchronous telerehabilitation group (Active Comparator)
  Interventions: Other: Synchronous exercise group

INTERVENTIONS:
Other: Asynchronous exercise group — Application of foot core training combined with lower extremity exercises using asynchronous telerehabilitation method.
  Arms: Asynchronous telerehabilitation group
Other: Synchronous exercise group — Application of foot core training combined with lower extremity exercises using synchronous telerehabilitation method.
  Arms: Synchronous telerehabilitation group

SUMMARY:
The aim of this study was to investigate the effects of lower extremity exercises combined with foot core exercise training on lower extremity pain, foot functionality, static and dynamic parameters of gait, and postural stability in individuals with rheumatoid arthritis using synchronous and asynchronous telerehabilitation methods.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with rheumatoid arthritis
* Being between the ages of 18-65
* Being willing to participate in the study

Exclusion Criteria:

* Having a neurological disease
* Having a pulmonary or cardiovascular problem that may affect daily life activities
* Sensory system disorders
* Having a history of surgery on the lower extremities or trunk
* Experiencing dizziness
* Having a cognitive disorder
* Having an additional rheumatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2025-10-24 (Estimated); Study Completion 2025-10-24 (Estimated)

PRIMARY OUTCOMES:
Foot Posture Index | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  It is a six-item index that determines foot posture. In this index, palpation of the distal talus medially and laterally, inequality in submalleolar and supramalleolar recesses, position of the calcaneus, medial protrusion of the navicular region in posterior observation, evaluation of the medial longitudinal arch, and the number of toes visible medially or laterally when viewed from the posterior will be evaluated. The examined regions are evaluated for each item up to (+2) according to the degree of pronation and up to (-2) according to the degree of supination, and the total score is obtained by summing these values.
Static Gait Analysis Evaluation | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  The evaluation will be made in a position where individuals stand with their arms free at their sides, their eyes fixed on a point 3 meters away in front, maintaining their posture as much as possible. In the static posture evaluation, the load on the right and left feet, and the right-left contact surface data will be evaluated and recorded. This parameter will be evaluated with the MultiSensor Platform 160 × 40 baropodometer device.
Dynamic Gait Analysis Evaluation | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  Individuals will be asked to walk at a speed they feel comfortable with, at least 8 steps on a 5-meter walking platform (3-meter platform and 2-meter walking analysis platform). The evaluation will be repeated 3 times. From the two-meter walking analysis 17 platform; left-right foot pressure percentage and left-right contact surfaces during walking will be obtained numerically and graphically. This parameter will be evaluated with the MultiSensor Platform 160 × 40 baropodometer device.
Postural Stability Assessment | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  Individuals will be asked to place their feet on the soles before measurements are taken, and the foot position of the individuals will not change during static measurements. For static load distribution measurement and bipedal balance measurement, individuals will be asked to keep their arms free next to their bodies and maintain their posture as much as possible by fixing their eyes on a point 3 meters in front. The measurement will be made with and without support, with eyes open and closed for 60 seconds. This parameter will be evaluated with the MultiSensor Platform 160 × 40 baropodometer device.

SECONDARY OUTCOMES:
Visual Analog Scale-Pain | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  Individuals' lower extremity and foot pain severity will be assessed using the Visual Analog Scale. Visual Analog Scale consisting of a single 100 mm line, used especially for pain assessment. The level of perceived negativity of the symptom increases as you move from left to right of the line. Individuals will be asked to make a mark on a horizontal or vertical line of 10 cm in length, starting with "I have no pain" and ending with "I have unbearable pain", where the severity of their pain will intersect this line. The distance from the lowest VAS level to the patient's mark will be measured with a ruler and recorded in centimeters.
Foot Function Index | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  The foot function index consists of 23 items with 3 subgroups: pain, disability and activity limitation. The pain subscale, which includes nine items, measures the level of foot pain in various situations, while the disability subscale, which includes nine items, determines the degree of difficulty in performing various functional activities due to foot problems. The activity limitation subscale, which includes five items, evaluates activity limitations due to foot problems. Patients score all items with the Visual Analog Scale (VAS), considering their foot conditions from the previous week. To calculate the subscales and the total score, the scores of each item are added, divided by the sum of the maximum scores of the items and multiplied by 100. Higher scores indicate more pain, disability and activity limitation. If the patient does not perform activities such as walking barefoot or using an orthosis, this item can be marked as not applicable and removed.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)